CLINICAL TRIAL: NCT00917215
Title: Effectiveness of Acupuncture for Asthma: A Randomized, Sham-acupuncture and Waiting-list Controlled Trial
Brief Title: Effectiveness of Acupuncture for Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea Institute of Oriental Medicine (Other Government)
Responsible Party: Sun-Mi Choi, Korea Institute of Oriental Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KE0802
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Asthma
Keywords: Asthma; Acupuncture; Pulmonary function; Quality of life
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- Active acupuncture (Experimental)
  Interventions: Device: Disposable stainless steel acupuncture (0.2mmx4mm)
- Sham acupuncture (Sham Comparator)
  Interventions: Device: Disposable stainless steel acupuncture (0.2mmx4mm)
- Waiting list control (No Intervention)

INTERVENTIONS:
Device: Disposable stainless steel acupuncture (0.2mmx4mm) — For active acupuncture group, needles were inserted into nine acupoints (CV22 and bilateral LU5, ST40, BL13, EXB1)with De-qi three times a week for 4 weeks.
  For sham acupuncture group, Nine non-acupoints corresponded with each active acupoint were treated with minimal penetration into skin three times a week for 4 weeks.
  Arms: Active acupuncture; Sham acupuncture

SUMMARY:
What is the trend of changes in asthmatic patients' daily peak expiratory flow (PEF) variability, pulmonary function, and quality of life (QOL) with acupuncture treatment on specific acupoints (CV22 and bilateral LU5, ST40, BL13, EXB1) compared with minimal acupuncture treatment (sham control group) on non-acupoints, and no acupuncture treatment (waiting list control group)?

ELIGIBILITY:
Inclusion Criteria:

* aged 19-70 years
* at least 12% improvement in forced expiratory volume in one second (FEV1)after the administration of short acting beta2 agonist.
* at least one typical asthmatic symptom
* using more than one routine anti-asthmatic medicine

Exclusion Criteria:

* acupuncture for asthma within 12 months of the study
* emergency department visit within one month of the study
* hospitalization for asthma within three months of the study
* severe upper respiratory tract infections within six weeks of the study
* systemic infections, cancers, autoimmune disorders, cardiac failures, myofacial infarcts,angina pectoris, renal failures or hepato-biliary diseases
* smoke more than ten cigarettes per day

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change of weekly average of peak expiratory flow (PEF)values in the morning at home | From 1 week of run-in period to the 4th week of treatment

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) Baseline Dyspnea Index (BDI) Transition Dyspnea Index (TDI) Quality of Life Questionnaire for Adult Korean Asthmatics (QLQAKA) | Baseline and 2 weeks, 4 weeks, 6 weeks after Baseline (BDI for baseline only, TDI for 2, 4, and 6 weeks after baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Allergy & Respiratory System, Department of Oriental Internal Medicine, Kyunghee medical center, Seoul, South Korea